CLINICAL TRIAL: NCT06455267
Title: A Single Center, Randomized Controlled Clinical Study on the Effect of L-ornithine on the Efficacy of Ustekinumab in Patients With Crohn's Disease
Brief Title: Preliminary Clinical Study on the Effect of L-ornithine on the Efficacy of Ustekinumab in Patients With Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ORN-XY3
Record Dates: First submitted 2024-05-23; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-04

CONDITIONS: Mild to Severe Crohns Disease
Keywords: Ustekinumab; L-ornithine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-ornithine supplementation group (Experimental): Patients in the L-ornithine supplementation group take oral ornithine capsules twice a day, three capsules per time, for 8 weeks, each containing 500mg of L-ornithine.
  Interventions: Dietary Supplement: Now Foods L-Ornithine Capsules
- control group (No Intervention): The control group did not receive additional intervention.

INTERVENTIONS:
Dietary Supplement: Now Foods L-Ornithine Capsules — L-ornithine is an amino acid that helps the liver clear toxic ammonia and plays an important role in liver protection and treatment of hepatic encephalopathy. Now Foods L-ornithine capsules are an ornithine supplement containing 500mg of L-ornithine per capsule. Patients in the L-ornithine supplementation group take ornithine capsules orally twice a day, three capsules each time, for 8 weeks.
  Arms: L-ornithine supplementation group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of supplementing L-ornithine compared to the control group on the efficacy of Ustekinumab in patients with Crohn's disease, and to summarize the role of supplementing L-ornithine in the treatment of CD patients.

Participants will be randomized into two groups: the L-ornithine supplementation group and the control group. The patients in the L-ornithine supplementation group received oral ornithine capsules for 8 weeks. The control group did not receive additional intervention. Follow up once a week, and after the study, patients will come to the hospital to finish the evaluation indicators.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effect of supplementing L-ornithine compared to the control group on the efficacy of Ustekinumab in patients with Crohn's disease, and to summarize the role of supplementing L-ornithine in the treatment of CD patients.

Participants will be randomized into two groups: the L-ornithine supplementation group and the control group. Patients in the L-ornithine supplementation group take oral ornithine capsules twice a day, three capsules per time, for 8 weeks, each containing 500mg of L-ornithine. The control group did not receive additional intervention. Follow up once a week, and after the study, patients will come to the hospital to finish the evaluation indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 75 years old;
2. Patients clinically diagnosed with Crohn's disease shall refer to the Chinese Guidelines for the Diagnosis and Treatment of Crohn's Disease (Guangzhou, 2023) for diagnostic criteria;
3. Patients receiving treatment with Ustekinumab;
4. Agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for inclusion in this study.

1. Patients with ALT or AST exceeding the normal upper limit by more than twice, and TBIL exceeding the normal upper limit by more than twice;
2. Patients with creatinine clearance rate less than 60ml/min;
3. Patients with severe active infections in the intestines or other areas that require the use of antibiotics or antiviral drugs;
4. Patients with intestinal tuberculosis, other chronic intestinal infectious diseases, and intestinal malignant tumors;
5. Pregnant and lactating women;
6. The fasting blood glucose of patients with diabetes or screening period exceeds 7.0mmol/L or glycosylated hemoglobin exceeds 6.5%;
7. Merge patients with severe mental illness, drug use, alcohol abuse, etc. who are unable to cooperate with the study;
8. Have participated in any other clinical research within the first month prior to enrollment;
9. The researcher determined that any other disease or condition is not suitable for patients participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Endoscopic remission rate | 8 weeks
  Endoscopic remission is defined using the Simple Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD score ranges from 0 to 60, where lower scores indicate less severe disease activity and higher scores indicate more severe disease activity. Endoscopic remission was defined as an SES-CD score ≤2.
Clinical remission rate | 8 weeks
  Clinical remission is defined using the Crohn's Disease Activity Index (CDAI). The CDAI score ranges from 0 to approximately 600, where lower scores indicate less severe disease activity and higher scores indicate more severe disease activity. Clinical remission was defined as a CDAI score ≤150.

SECONDARY OUTCOMES:
Biomarker target attainment rate | 8 weeks
  The target of inflammatory biomarkers is defined using the following scales:
  * C-Reactive Protein (CRP): CRP levels less than 5 mg/L. The CRP scale ranges from 0 to >100 mg/L, with higher scores indicating higher levels of inflammation.
  * Erythrocyte Sedimentation Rate (ESR): ESR levels less than 15 mm/hr for men and less than 20 mm/hr for women. The ESR scale ranges from 0 to >100 mm/hr, with higher scores indicating higher levels of inflammation.
  * Fecal Calprotectin (FC): FC levels decreased to 100-250 µg/g. The FC scale ranges from 0 to >500 µg/g, with higher scores indicating higher levels of intestinal inflammation.
  The biomarker target attainment rate is the percentage of patients who meet all three criteria at the end of the 8-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University; Jie Hong, PHD, Principal Investigator — RenJi Hospital
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Some data underlying this trial cannot be shared publicly due to protection of participant's privacy.